CLINICAL TRIAL: NCT02291484
Title: Comprehensive Cardiac CT Versus Exercise Testing in Suspected Coronary Artery Disease (2)
Acronym: CRESCENT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Koen Nieman, Dr K Nieman, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC2013022
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Stable Angina Pectoris; Coronary Artery Disease
Keywords: Computed tomography; Coronary angiography; Coronary artery disease; Perfusion imaging; Comparative effectiveness; Randomized controlled trial; Cost-effectiveness
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive cardiac CT (Experimental): Tiered cardiac CT protocol:
  1. CT calcium scan
  2. CT angiography (if calcium scan positive or high pre-test probability)
  3. CT perfusion (if >50% stenosis on CTA, or cannot be ruled out)
  Interventions: Device: Cardiac CT scan
- Standard care (No Intervention): Standard diagnostic management of suspected CAD, using stress testing

INTERVENTIONS:
Device: Cardiac CT scan — CT-guided management
  Arms: Comprehensive cardiac CT

SUMMARY:
Multi-center, randomized-controlled trial comparing a comprehensive cardiac CT protocol with standard stress testing in patients with stable chest pain complaints.

DETAILED DESCRIPTION:
Rationale: CT calcium and coronary lumen imaging allow efficient exclusion of coronary artery disease (CAD), but cannot assess the hemodynamic significance of obstructive findings. Addition of stress myocardial perfusion imaging, which assesses the functional relevance of coronary narrowing, completes the non-invasive cardiac evaluation.

Hypothesis: A comprehensive cardiac CT examination will allow fast, accurate and complete evaluation of suspected CAD.

Objective: evaluate the effectiveness and efficiency of comprehensive cardiac CT workup of suspected CAD.

Study design: Open-labelled, randomized-controlled, clinical efficiency trial, with an intention-to-diagnose approach, between CT-guided management and the current standard of care (based on functional testing of provocable myocardial ischemia) in patients with suspected CAD.

Study population: 250 patients (>18 yrs) with stable chest complaints, a >10% pre-test probability of CAD, and referred for evaluation of possible CAD.

Intervention: Instead of the usual diagnostic approach, patients in the intervention group will undergo in sequence the following CT examinations: coronary calcium scan, coronary CT angiography and CT myocardial perfusion imaging, with completion dependent on results. Findings on CT will direct further management.

Main study parameters/endpoints:

Primary: Rate of negative invasive angiograms (as percentage of total population) Secondary: Diagnostic yield, chest complaints, quality of life, diagnostic and therapeutic procedures, overall costs and adverse events at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years.
* Chest pain symptoms suspicious of coronary heart disease.
* Pre-test probability of coronary artery disease >10%

Exclusion Criteria:

* History of CAD: prior myocardial infarction or revascularization procedure
* Contra-indication to radiation exposure (CT/SPECT): pregnancy
* Contra-indication to iodine contrast media: renal failure, iodine allergy
* Contra-indications to adenosine
* Inability or unwillingness to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of negative invasive angiograms (as percentage of total population) | 6 months
  Number of performed invasive angiograms with no CAD requiring intervention

SECONDARY OUTCOMES:
Chest pain complaints | 6 months
  Proportion of patients experiencing symptoms of chest pain
Quality of life | 6 months
  Questionnaire based quality of life score
Major adverse event rate | 6 months
  Death, myocardial infarction, unstable angina, urgent revascularizations, CVA
Radiation exposure | 6 months
  Cumulative radiation dose from diagnostic and therapeutic interventions
Number of diagnostic and therapeutic procedures | 6 months
  Number of diagnostic and therapeutic procedures
Medical expenses | 6 months
  All medical expenses related to the diagnosis and treatment of suspected CAD

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - Albert Schweizerzieknhuis, Dordrecht
  - Maastricht University Medical Center, Maastricht
  - Erasmus MC, Rotterdam
  - Maasstadziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lubbers M, Coenen A, Kofflard M, Bruning T, Kietselaer B, Galema T, Kock M, Niezen A, Das M, van Gent M, van den Bos EJ, van Woerkens L, Musters P, Kooij S, Nous F, Budde R, Hunink M, Nieman K. Comprehensive Cardiac CT With Myocardial Perfusion Imaging Versus Functional Testing in Suspected Coronary Artery Disease: The Multicenter, Randomized CRESCENT-II Trial. JACC Cardiovasc Imaging. 2018 Nov;11(11):1625-1636. doi: 10.1016/j.jcmg.2017.10.010. Epub 2017 Dec 13. PMID 29248657